CLINICAL TRIAL: NCT05845892
Title: EFFECT OF STRESS BALL ON COMFORT AND ANXIETY IN HEMODIALYSIS PATIENTS: RANDOMIZED CONTROLLED TRIAL
Brief Title: EFFECT OF STRESS BALL ON COMFORT AND ANXIETY CONTROLLED TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevil Şahin, Assoc Prof Dr, TC Erciyes University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/740
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Anxiety; Comfort
Keywords: hemodialysis, comfort, anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: With this randomized controlled trial, it is aimed to determine the anxiety levels and comfort levels of the patients by using a total of 30 minutes of stress ball at the beginning and during 9 sessions of hemodialysis treatment in patients receiving hemodialysis treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will be given written and oral consent by explaining the purpose of the study. Patients with fistula and non-grafted arms will be asked to fill out data collection forms at the first interview. Patients will then be asked to squeeze the stress ball 15 minutes before the start of hemodialysis treatment and for 15 minutes during hemodialysis treatment. This treatment will be performed during (nine) hemodialysis treatments. After the last session, data collection forms will be filled out again.
  Use of stress Ball
  1) place a stress ball in one hand (which hand will be left to the patients' wishes.) 2.squeeze the ball in your hand for 2-3 seconds after receiving it and then loosen it.
  3.perform this application for a total of 30 minutes before and during hemodialysis treatment.
  Interventions: Other: stress ball
- Control (No Intervention): No intervention will be given to the control group other than standard treatment. Data collection forms will be completed before the first dialysis session and after the eighth session.
  Before the first dialysis session and after the ninth session, the individual Introduction form, the Visual Analog scale (VAS) for stress level, the Beck anxiety scale and the hemodialysis comfort scale will be filled out.

INTERVENTIONS:
Other: stress ball — The use of the stress ball by the experimental group patients will be reminded by a hemodialysis nurse who was not involved in the study.
  Arms: Intervention

SUMMARY:
In this study, it was aimed to determine the anxiety levels and comfort levels of the patients using stress ball in patients receiving hemodialysis treatment.

This study was conducted as a randomized controlled trial. The universe of the study consisted of 156 patients receiving HD treatment at a special hemodialysis center. The study was completed with a total of 63 patients, including 31 people in the intervention group and 32 people in the control group, who met the criteria for inclusion in the study between 27.02.2023 and 27.03.2023.

The individual demonstration form was used to collect data, the Visual Analog scale (VAS) for stress level and the hemodialysis comfort scale.

DETAILED DESCRIPTION:
Procedures administered to intervention groups:

Patients will be given written and oral consent by explaining the purpose of the study. Patients with fistula and non-grafted arms will be asked to fill out data collection forms at the first interview. Patients will then be asked to squeeze the stress ball 15 minutes before the start of hemodialysis treatment and for 15 minutes during hemodialysis treatment. This treatment will be performed during the 9 (nine) hemodialysis treatment. After the last session, data collection forms will be filled out again.

Use of stress Ball

1) Place a stress ball in one hand (which hand will be left to the patients' wishes.) 2.Squeeze the ball in your hand for 2-3 seconds after receiving it and then loosen it.

3.Perform this application for a total of 30 minutes before and during hemodialysis treatment.

Procedures administered to control groups:

No intervention will be given to the control group other than standard treatment. Data collection forms will be completed before the first dialysis session and after the ninth session.

ELIGIBILITY:
Inclusion Criteria:

* Who is over 18 years old
* Having been on an average of four hours of hemodialysis program, three times a week, for at least 6 months;
* Who can respond in writing or verbally to the scales applied,
* In addition to last-stage kidney disease, there is no physical deficiency,
* Can apply stress ball as shown during hemodialysis work
* Individuals who agree to participate in the research

Exclusion Criteria:

* With fistula on both arms
* People with psychiatric problems
* With nerve, soft tissue and vascular disease in the upper extremity
* Out of town during work

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Scale | One mounth.
  Developed by Beck et al. (1988). The Cronbach alpha coefficient of the original scale is .93. The Turkish version of the Beck anxiety scale was prepared by Ulusoy et al. (1998). The scale consists of 21 items and two sub-dimensions.
  BAO provides quadruple lycert-type measurement. The lowest possible score on the scale is 0 and the highest score is 63. Those who answered "never" to the scale questions received 0 points, those who answered "it did not affect much at a light level" received 1 points, those who answered "it was not pleasant, but I was able to endure" received 2 points, and those who answered "on a serious level, I was very hard to endure" received 3 points. The total score on the scale indicates

SECONDARY OUTCOMES:
Hemodialysis Comfort Scale | One mounth
  The General comfort scale developed by Kolcaba and the comfort scales developed specific to certain situations after it is a scale of the five likert type, which was validated and trusted by Şahin-Orak and his colleagues in 2017, consists of 9 items and 2 sub-dimensions. At least 3.00 and at most 15.00 points can be taken from the relaxation sub-dimension; at least 7.00 and at most 30.00 points can be taken from the overcoming sub-dimension. The lowest score from HDKO is 9, the highest score is 45. As the score gets closer to 45, the comfort level incre

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes Universty, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan